CLINICAL TRIAL: NCT04363034
Title: Arkansas Expanded Access COVID-19 Convalescent Plasma Treatment Program
Status: No longer available | Type: Expanded Access
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 260944
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: Convalescent Plasma — 1-2 units (200-400 mL per unit, not to exceed 550 mL total) of ABO compatible, low isohemagglutinin titer, COVID-19 convalescent plasma

SUMMARY:
This is an expanded access treatment protocol to treat up to 100 patients with severe or life-threatening, laboratory confirmed COVID-19 with COVID-19 convalescent plasma.

DETAILED DESCRIPTION:
This is an expanded access treatment protocol to treat up to 100 subjects with severe or life-threatening, laboratory confirmed COVID-19 with COVID-19 convalescent plasma. Subjects will receive 1-2 units (200-400 mL per unit, not to exceed 550 mL total) of ABO compatible, low isohemagglutinin titer, COVID-19 convalescent plasma. Plasma will be administered one unit per day for up to two days. The duration of infusion will usually take 1 to 2 hours (rate of 100 to 250 mL/hr). The infusion should not exceed 4 hours. Plasma infusions will be administered following standard institutional procedures, including the use of premedications (e.g. acetaminophen, diphenhydramine, etc.) as necessary.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* 18 years of age or older
* Laboratory confirmed COVID-19 via SARS-CoV-2 RT-PCR testing
* Patients currently hospitalized with severe or life-threatening COVID-19 or patients the treating physician deems to be at high-risk for progressing to severe or life-threatening COVID-19.

  * Severe disease, defined as one or more of the following:

    * dyspnea,
    * respiratory frequency ≥ 30/min,
    * blood oxygen saturation ≤ 93%,
    * partial pressure of arterial oxygen to fraction of inspired oxygen ratio < 300, and/or
    * lung infiltrates > 50% within 24 to 48 hours
  * Life-threatening disease, defined as one or more of the following:

    * respiratory failure,
    * septic shock, and/or
    * multiple organ dysfunction or failure
* Patients or their legally authorized representative must provide informed consent.

Exclusion Criteria:

* Female patients with positive pregnancy test, breastfeeding, or planning to become pregnant/breastfeed during the study period.
* Patients who have received pooled immunoglobulin in past 30 days
* Contraindication to transfusions or history of prior reactions to transfusion blood products

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult